CLINICAL TRIAL: NCT02647177
Title: A Prospective Study To Identify Predictive Biological Markers In Blood And Cyst Fluid Aspirates From Patients With Pancreatic Cyst Lesions
Status: Recruiting | Type: Observational
Sponsor: The University of Texas Health Science Center, Houston (Other)
Responsible Party: Principal Investigator, Nirav C Thosani, Assistant Professor, The University of Texas Health Science Center, Houston
Other Study IDs: HSC-MS-14-0980
Record Dates: First submitted 2016-01-04; First posted 2016-01-06 (Estimated); Last update posted 2025-08-15 (Actual); Status verified 2025-08

CONDITIONS: Pancreatic Cystic Lesions

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Cross-Sectional
Patient Registry: Yes
Target Follow-Up Duration: 1 Year
Biospecimen Retention: Samples With DNA — Cyst aspirate
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Pancreatic Cyst Group: Only the eligible participant in the study are considered for inclusion in this group.
  Interventions: Other: Pancreatic Cyst Aspiration

INTERVENTIONS:
Other: Pancreatic Cyst Aspiration — 10 CC of pancreatic cyst aspiration

SUMMARY:
The purpose To determine the diagnostic potential of various biological markers in blood and cyst fluid aspirates from patients with Pancreatic Cystic Lesions (PCLs).

Research design This is a 10-year prospective cohort and pancreatic cyst fluid repository study enrolling all patients diagnosed with pancreatic cyst and undergoing the cyst aspiration.

Procedures to be used Blood Sample Cyst Fluid Sample

Data Collection:

Medical Record Number Demographics (age, sex, gender, race) Contact information History of alcohol use and IV and other recreational drugs and narcotics use/abuse Medication history Past hospitalizations, diagnoses, and treatment Physical examination findings Imaging data of abdominal and chest regions, including and not limited to ultrasonography, magnetic resonance imaging (MRI), computed tomography (CT) Future admissions, diagnoses, treatment including histopathological findings of resected specimens and blood reports End of study data: clinical progression of disease, cyst size, wall thickening, calcification, communication with pancreatic duct, string sign, cytology, immunohistochemical findings, assay levels of lipase, amylase CEA (carcinoembryonic antigen), carbohydrate antigen19-9 (CA 19-9), and other biomarkers.

Risks and potential benefits The risks associated with this study are slight discomfort or bruising from the blood sampling and the possible loss of confidentiality if the patient data or information is inadvertently disclosed outside of this study. The patient will not receive any additional benefit from the study aside from those received as part of routine standard of care.

Importance of knowledge that may reasonably be expected to result The knowledge gained from this study may benefit other patients with Pancreatic Cyst Lesions in the future.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of Pancreatic Cystic Lesions (PCLs) or Acute Pancreatitis (AP) or chronic pancreatitis(CP) or Pancreatic Cancer (PC) (any stage/grade) or congenital developmental anomalies of the pancreas.
* Any combination of the diagnoses above.
* Patients must provide written informed consent for the collection of blood specimens for research purposes.
* Patients with PCLs must provide informed consent for collection of excess cyst fluid aspirate remaining after testing for routine standard of care
* Patients with pancreatic Cystic Lesions (PCLs) or AP or CP or PC (any stage/grade) or congenital developmental anomalies of the pancreas undergoing surgery must provide informed consent for collection of surgical specimen

Exclusion Criteria:

* Patients with co-existing malignancies of other organs (or prior history of such)
* Patients unable to provide informed consent
* Patients unable to complete follow up

Ages: 18 Years to 100 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients presenting to Memorial Hermann Hospital for care with the primary and subinvestigator(s) of the study will be identified, prescreened for eligibility and listed for informed consent and subsequent enrollment.
Sampling Method: Non-Probability Sample
Enrollment: 1000 (Estimated)
Dates: Start 2015-05 (Actual); Primary Completion 2027-04 (Estimated); Study Completion 2027-04 (Estimated)

PRIMARY OUTCOMES:
Detection of early progression to Tumor | 2 years
  To identify any correlation between higher expression levels with early progression to malignant changes in the pancreas

CONTACTS AND LOCATIONS:
Overall Officials: Nirav C Thosani, MD MHA, Principal Investigator — The University of Texas Health Science Center, Houston
Locations (1):
- The University of Texas Health Science Center at Houston, Houston, Texas, United States